CLINICAL TRIAL: NCT07116824
Title: A Phase II Trial to Evaluate the Safety and Efficacy of HB1801 Combination Therapy as First-line Treatment in HER2-positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: HB1801 Combined Treatment of HER2-positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-014
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab; pertuzumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-center, randomized, Phase II clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1：Combination of HB1801, Trastuzumab and Pertuzumab (Experimental): HB1801: per protocol; Trastuzumab: 8mg/kg loading dose and then 6mg/kg, Q3W; Pertuzumab: 840mg loading dose and then 420mg, Q3W
  Interventions: Drug: HB1801; Drug: Trastuzumab; Drug: Pertuzumab
- Cohort 2：Combination of Docetaxel, Trastuzumab and Pertuzumab (Active Comparator): Docetaxel：75mg/m^2 ，Q3W Trastuzumab: 8mg/kg loading dose and then 6mg/kg, Q3W; Pertuzumab: 840mg loading dose and then 420mg, Q3W
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: HB1801 — HB1801 is administered by intravenous infusion.
  Arms: Cohort 1：Combination of HB1801, Trastuzumab and Pertuzumab
Drug: Trastuzumab — Trastuzumab is administered by intravenous infusion, 8mg/kg loading dose and then 6mg/kg per cycle, Q3W.
Drug: Pertuzumab — Pertuzumab is administered by intravenous infusion, 840mg loading dose and then 420mg per cycle, Q3W.
Drug: Docetaxel — Docetaxel is administered by intravenous infusion, 75mg/m^2, Q3W.
  Arms: Cohort 2：Combination of Docetaxel, Trastuzumab and Pertuzumab

SUMMARY:
This study is designed to evaluate the safety and efficacy of HB1801 combination therapy as first-line treatment in HER2-positive unresectable locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study and sign the Informed Consent Form (ICF);
* Age ≥ 18 years;
* Histologically and/or cytologically confirmed unresectable locally recurrent or metastatic breast cancer;
* HER2-positive (IHC 3+, or IHC 2+ with ISH-positive);
* No prior systemic chemotherapy and/or HER2-targeted therapy for unresectable locally recurrent or metastatic breast cancer (participants who have received ≤1 line of endocrine therapy are eligible); Participants who relapsed >12 months after completing (neo)adjuvant chemotherapy or HER2-targeted therapy may be considered for enrollment;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* At least one measurable lesion per RECIST 1.1. The measurable lesion should not have received local treatment such as radiotherapy (lesions in previously irradiated areas may be selected as target lesions if progression is confirmed). Target lesions cannot be bone-only metastases;
* Adequate organ and bone marrow function (without transfusion or hematopoietic growth factor support within 14 days prior to testing):

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
  2. Platelet count ≥ 100 × 10^9/L;
  3. Hemoglobin ≥ 90 g/L;
  4. Liver function: Total bilirubin (TBIL) ≤ 1.0 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (ALT/AST≤ 5 × ULN for participants with liver metastases; AST/ALT ≤ 1.5 × ULN for participants with alkaline phosphatase (ALP) > 2.5 × ULN);
  5. Renal function: Creatinine clearance ≥60 mL/min (calculated by Cockcroft-Gault formula);
  6. Coagulation: International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (for participants receiving anticoagulation therapy, the investigator should confirm that INR and APTT are within safe and effective therapeutic ranges);
  7. Left ventricular ejection fraction (LVEF) > 50%;
* Expected survival ≥ 3 months;
* For women of childbearing potential: Negative serum pregnancy test within 7 days before randomization and agreement to use reliable contraception during the study and for 3 months after last dose of docetaxel/HB1801 or 7 months after last dose of trastuzumab/pertuzumab (whichever is longer). For male participants with partners of childbearing potential: Agreement to use reliable contraception during the study and for 3 months after last dose of docetaxel/HB1801 or 7 months after last dose of trastuzumab/pertuzumab (whichever is longer).

Exclusion Criteria:

* Contraindications to trastuzumab, pertuzumab, or docetaxel, or deemed by the investigator as unsuitable for treatment with HB1801, docetaxel, pertuzumab, or trastuzumab;
* Participants with ≥ Grade 3 peripheral neuropathy at randomization;
* Toxicities from prior anticancer therapy have not resolved to ≤ Grade 1 per CTCAE v5.0 (except for alopecia, peripheral neuropathy, or laboratory abnormalities deemed non-risky by the investigator, which must be ≤ Grade 2);
* History of LVEF decline to < 50%, symptomatic congestive heart failure (CHF), or toxicity leading to permanent discontinuation during prior HER2-targeted therapy;
* Known hypersensitivity or contraindications to corticosteroids (including but not limited to active peptic ulcer, severe hypertension, severe hypokalemia, glaucoma, etc.);
* Prior anthracycline therapy exceeding cumulative doses of: Doxorubicin or liposomal doxorubicin > 360 mg/m², Epirubicin > 720 mg/m², Mitoxantrone > 120 mg/m², Other anthracyclines > doxorubicin-equivalent 360 mg/m²(If multiple anthracyclines were used, the total dose must not exceed 360 mg/m² doxorubicin-equivalent);
* Use of strong CYP3A4 inhibitors within 14 days before randomization;
* History of hypersensitivity to any study drug component or excipients;
* Untreated or unstable brain/spinal metastases, leptomeningeal disease, or cord compression (participants with treated, asymptomatic CNS lesions stable for ≥4 weeks on imaging, without edema, and off corticosteroids may be eligible);
* Active malignancies within 3 years prior to randomization, except: studied breast cancer, locally cured tumors (e.g., resected basal/squamous skin cancer, superficial bladder cancer, cervical/breast carcinoma in situ, early-stage thyroid cancer);
* Uncontrolled or significant cardiovascular disease, including:

  1. NYHA Class II+ CHF, unstable angina, myocardial infarction, or hemodynamically unstable arrhythmia within 6 months;
  2. Primary cardiomyopathy (e.g., dilated, hypertrophic, arrhythmogenic right ventricular, restrictive);
  3. Clinically significant QTc prolongation (Fridericia-corrected QTcF > 450 ms at screening);
  4. Arterial/venous thromboembolism within 6 months (e.g., stroke, TIA, DVT, PE);
  5. Uncontrolled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg);
* Active/chronic infection requiring systemic antimicrobial/antiviral therapy within 14 days (including tuberculosis);
* Active hepatitis: HBV (HBsAg+ with HBV-DNA ≥ 2×10³ IU/mL), HCV (anti-HCV+ with detectable HCV-RNA) *Note: HBsAg+ carriers with HBV-DNA < 2×10³ IU/mL may enroll if willing to receive entecavir/antiviral therapy;*
* Known HIV infection;
* Concurrent participation in other interventional clinical trials (except observational studies or follow-up phases) or <4 weeks since last dose in prior interventional trials;
* Anticancer therapy within 28 days (radiotherapy, targeted/immunotherapy, investigational drugs) or 14 days (traditional Chinese medicine with antitumor indications);
* Uncontrolled effusions requiring frequent drainage/medical intervention within 7 days (e.g., pleural, ascites, pericardial) or needing re-intervention within 2 weeks (excluding cytology);
* Major surgery within 28 days (excluding biopsies);
* Pregnant or lactating women;
* Other conditions compromising study participation/benefit (e.g., psychiatric disorders, substance abuse, or clinically significant comorbidities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-11-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as assessed by RECIST 1.1 | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) as assessed by RECIST 1.1 | Up to approximately 2 years
Duration of Response (DoR) as assessed by RECIST 1.1 | Up to approximately 2 years
Progression-free survival (PFS) as assessed by RECIST 1.1 | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 2 years
Incidence and severity of treatment-emergent adverse events (TEAE) | Up to approximately 2 years